CLINICAL TRIAL: NCT01439100
Title: A Randomised Placebo Controlled Study of OXN PR for Severe Parkinson's Disease Associated Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OXN2504; 2011-002901-31 (EudraCT Number)
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease With Severe Pain
Keywords: Parkinson's disease; severe pain; OXN PR; randomised
MeSH Terms: conditions — Parkinson Disease; Pain | interventions — Oxycodone

ARMS (2):
- OXN PR (Active Comparator): Oxycodone/Naloxone Prolonged Release tablets
  Interventions: Drug: Oxycodone/Naloxone Prolonged Release tablets
- Dummy tablet (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone/Naloxone Prolonged Release tablets
  Arms: OXN PR
Drug: Placebo — Dummy tablet
  Arms: Dummy tablet

SUMMARY:
To demonstrate superiority of OXN PR compared to placebo with respect to analgesic efficacy in subjects with chronic severe pain associated with Parkinson's disease (PD), as assessed by averaged 24 hour pain scores collected for 7 days prior to the clinic visits

DETAILED DESCRIPTION:
Pain management in PD is a recognised unmet need. Estimates of incidence vary in the literature from 29% to 83%. The types and sources of pain experienced by PD patients vary and include: musculoskeletal pain, PD related chronic pain, fluctuation-related pain, nocturnal pain, coat-hanger pain, oro-facial pain and peripheral limb or abdominal pain (also including drug-induced pain). Whilst modifications to dosing of dopaminergic therapy represents the most common method of controlling some of these pain symptoms, this must be balanced against the worsening of side effects of increased doses of this treatment type.

Oxycodone hydrochloride and naloxone hydrochloride dihydrate combined oral prolonged release tablets (OXN PR), is the investigational product to be used in this study. OXN PR is a prolonged release tablet consisting of oxycodone and naloxone in a 2:1 ratio. Due to the local competitive antagonism of the opioid receptor-mediated oxycodone effect by naloxone in the gut, naloxone reduces opioid-associated bowel dysfunction.

The purpose of this study is to investigate whether effective pain control for the treatment of PD associated pain may be achieved with OXN PR. The secondary considerations for this study are to examine whether OXN PR may offer any additional benefits to the patients Quality of Life or symptoms of PD. If effective pain relief can be achieved with an analgesic without the side effects described in above, this could reduce the need to increase the dose of dopaminergic medications to manage pain, and therefore reduce the negative side effects of dopaminergic therapy described above. Given the prevalence of constipation in this patient population the bowel sparing effects of the OXN PR combination treatment may provide an ethical rationale for its use over that of other opioids.

ELIGIBILITY:
Inclusion Criteria

1. Males and females, age of 25 years or over
2. Able to provide written informed consent
3. Primary diagnosis of Parkinson's disease Stage II-IV)
4. Graded as having severe pain
5. An average pain score of 6 or above on an 11 point NRS, over the previous 7 days
6. Female subjects willing to use an adequate and highly effective method of contraception throughout the study.
7. Subjects likely to benefit from WHO step III opioid therapy for the duration of the study
8. Subjects must not have received opioid containing medication in the last 6 months on a regular basis
9. Receiving stable treatment for Parkinson's disease for at least 4 weeks prior to randomisation
10. Subject does not have visual or auditory impairments that would reduce their ability to complete study questionnaires or be unable to receive instructions for these
11. Concomitant medication (including co-analgesic) use anticipated to remain stable throughout the Double-Blind Phase of the study
12. Subjects willing and able to participate in all aspects of the study and comply with the use of study medication.

Open-Label Extension Inclusion Criteria

The aim of the Open-Label Phase is to ensure a safe transfer of all subjects to a subsequent pain treatment after the study. Subjects must:

1. Still meet general inclusion criteria for Double-Blind Phase; subjects do not have to meet inclusion 5, 6, 9 & 12
2. Have completed the Double-Blind Phase or discontinued early but have had at least 8 weeks treatment with study medication.

Exclusion Criteria

Subjects who are to be excluded from the study are those who meet any of the following criteria:

Medical Conditions

1. Cognitive impairment as assessed with the MMSE scoring 24 or less
2. History of psychosis (hallucinations, delusions, etc.)
3. History of drug or alcohol abuse or current compulsive addictive use of drugs or alcohol
4. Parkinsonian-like disease secondary to drug therapy side-effects e.g. due to exposure to medications that deplete dopamine (reserpine, tetrabenazine) or block dopamine receptors (neuroleptics, antiemetics)
5. Parkinson-plus syndromes e.g. progressive supranuclear palsy (PSP) and the multiple system atrophies (MSA)
6. Females who are pregnant (positive β-hCG test) or lactating
7. Any other contraindications to use of the opioid study medication(s) as per the SmPC/IB:

   * Hypersensitivity to the active substances or to any of the excipients
   * Any situation where opioids are contraindicated
   * Severe respiratory depression with hypoxia and/or hypercapnia
   * Severe chronic obstructive pulmonary disease
   * Cor pulmonal
   * Severe bronchial asthma
   * Non-opioid induced paralytic ileus
   * Moderate to severe hepatic impairment (see exclusion criterion 16)
8. Any other contraindications to use of the study Double-Blind Phase rescue medication as per the SmPC:

   * known hypersensitivity to levodopa or benserazide
   * contra-indicated in narrow-angle glaucoma (it may be used in wide-angle glaucoma provided that the intra-ocular pressure remains under control); severe psychoneuroses or psychoses; severe endocrine, renal, hepatic or cardiac disorders
   * should not be given in conjunction with, or within 2 weeks of withdrawal of, monoamine oxidase (MAO) inhibitors, except selective MAO-B inhibitors (e.g. selegiline) or selective MAO-A inhibitors (e.g. moclobemide) unless selective MAO inhibitors are given in combination in which case it is contraindicated
   * not be used in persons who have a history of, or who may be suffering from, a malignant melanoma
9. Subjects with any of the following as determined by medical history, clinical laboratory tests, ECG results, and physical examination, that would place the subject at risk upon exposure to the study medication:

   * myxoedema
   * untreated hypothyroidism
   * Addison's disease
   * increase of intracranial pressure
   * uncontrolled seizures or convulsive disorder
   * evidence of clinically significant cardiovascular, renal, hepatic, gastrointestinal (e.g. paralytic ileus), or psychiatric disease (subjects with controlled co-morbidities may be included following agreement with the Medical Monitor) Contraindicated Treatments
10. Treatment with Deep Brain Stimulation
11. Subjects receiving hypnotics or other central nervous system (CNS) depressants that, in the Investigator's opinion, may pose a risk of additional CNS depression with opioids study medication
12. Subjects presently taking, or who have taken, naloxone or naltrexone less than or equal to 30 days prior to the Screening Visit
13. Subjects who have received an investigational medicinal product within 30 days of study entry (defined as the start of the Screening Phase)
14. Any current use of an opioid other than the study medication provided
15. Subjects with a positive urine drug test at Screening Visit 1, which indicates unreported illicit drug use or unreported use of a concomitant medication not required to treat the Subjects' medical condition(s) Laboratory Exclusions
16. Abnormal parameters as defined:

    * aspartate aminotransferase (AST; SGOT) > 3 times the upper limit of normal
    * alanine aminotransferase (ALT; SGPT) > 3 times the upper limit of normal
    * alkaline phosphatase levels > 3 times the upper limit of normal
    * gamma glutamyl transpeptidase (GGT or GGTP) > 3 times the upper limit of normal
    * Abnormal total bilirubin and/or creatinine level(s) > 1.5 times the upper limit of normal. Subjects whose total bilirubin levels or creatinine levels are below the lower limit of normal can participate in the study if they meet the criteria below:

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- Czechia (5):
  - Fakultní nemocnice u sv. Anny v Brně Neurologická klinika, Brno
  - Poliklinika Choceň Neuroligická ambulance, Choceň
  - Fakultní nemocnice Plzeň Neurologická klinika, Plzeň-Lochotín
  - Neurologická ambulance, Polička
  - CTC Rychnov nad Kněžnou s.r.o., Rychnov nad Kněžnou
- Germany (9):
  - Ruhr Universität Bochum St. Josef-Hospital, Bochum
  - Universitätsmedizin Göttingen Georg-August-Universität, Göttingen
  - Zentrum für Altersmedizin, Haag I. OB
  - Paracelsus-Elena-Klinik, Kassel
  - Uniklinik Leipzig, Leipzig
  - Philipps-Universität, Marburg
  - Asklepios Fachklinikum Abteilung für Neurologie, Stadtroda
  - Neurologie Berlin, Steglitz
  - Uniklinik Ulm, Ulm
- Hungary (6):
  - Szent János Kórháza és Észak-budai Egyesített Kórházaik, Budapest
  - Kenézy Kórház-Rendelőintézet Egészségügyi Szolgáltató Kft., Debrecen
  - Szent Pantaleon Kórház-Rendelőintézet Dunaújváros, Dunaújváros
  - Vaszary Kolos Kórház Esztergom, Esztergom
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Bács-Kiskun Megyei Kórháza, Kecskemét
- Poland (2):
  - NZOZ Synapsa, Kielce
  - Krakowska Akademia Neurologii Sp. z o.o., Krakow
- Spitalul Clinic de Neuropsihiatrie, Craiova, Jud. Dolj, Romania
- Spain (4):
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - USP Institut Universitari Dexeus, Barcelona
  - Hospital Universtario La Paz, Madrid
  - Hospital General de Catalunya, Sant Cugat, Barcelona
- United Kingdom (4):
  - Fairfield General Hospital Pennine Acute NHS Trust, Bury Great Manchester
  - King's College Hospital NHS Foundation Trust, London
  - Royal Preston Hospital, Preston
  - City General Hospital, Pharmacy Dept, Newcastle Road, Stoke-on-Trent

REFERENCES:
- [Derived] Trenkwalder C, Chaudhuri KR, Martinez-Martin P, Rascol O, Ehret R, Valis M, Satori M, Krygowska-Wajs A, Marti MJ, Reimer K, Oksche A, Lomax M, DeCesare J, Hopp M; PANDA study group. Prolonged-release oxycodone-naloxone for treatment of severe pain in patients with Parkinson's disease (PANDA): a double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2015 Dec;14(12):1161-70. doi: 10.1016/S1474-4422(15)00243-4. Epub 2015 Oct 19. PMID 26494524